CLINICAL TRIAL: NCT01261481
Title: Comparison of the Relative Oral Bioavailability of Tolvaptan Administered Via Nasogastric Tube to Tolvaptan Tablets Swallowed Intact
Brief Title: Bioavailability Study Comparing Tolvaptan Administered Via Nasogastric Tube to Tolvaptan Tablets Swallowed Intact
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Otsuka America Pharmaceutical (Industry)
Responsible Party: Principal Investigator, Herb Patterson, PharmD, Professor and Executive Vice Chair, DPET, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 10-1865
Record Dates: First submitted 2010-12-14; First posted 2010-12-16 (Estimated); Last update posted 2012-12-07 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Bioavailability
MeSH Terms: interventions — Tolvaptan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tolvaptan Intact Tablet Orally (Experimental)
  Interventions: Drug: Tolvaptan
- Tolvaptan via Nasogastric Tube (Experimental)
  Interventions: Drug: Tolvaptan

INTERVENTIONS:
Drug: Tolvaptan — Tolvaptan 15 mg administered once orally as an intact tablet.
  Other Names: Samsca
  Arms: Tolvaptan Intact Tablet Orally
Drug: Tolvaptan — Tolvaptan 15 mg administered once via nasogastric tube.
  Other Names: Samsca
  Arms: Tolvaptan via Nasogastric Tube

SUMMARY:
The purpose of the study is to compare the relative bioavailability and pharmacokinetics of tolvaptan 15 mg tablets administered orally versus tolvaptan via nasogastric (NG) tube in healthy male and female subjects.

This study is an open 2-treatment, 2-period, 2-sequence crossover study to compare the relative bioavailability of tolvaptan tablets to tolvaptan given via nasogastric tube in 28 healthy adults. Subjects will be randomized to one of the two treatment sequences; either tolvaptan oral tablets swallowed intact followed by a tablet crushed and administered via nasogastric tube, or the reverse sequence. Serial pharmacokinetic samples will be collected following each tolvaptan administration and safety assessments will be performed. The relative bioavailability of tolvaptan administered via nasogastric tube will be compared to tolvaptan tablets swallowed intact.

DETAILED DESCRIPTION:
This study is an open 2-treatment, 2-period, 2-sequence crossover study to compare the relative bioavailability of tolvaptan tablets to tolvaptan NG in 28 healthy adults. The study will be conducted at the University of North Carolina (UNC) Hospital in the Clinical Translational Research Center (CTRC). The study will consist of three phases (screening and two drug administration visits). Subjects will be randomized to one of the two treatment sequences; either tolvaptan oral tablets swallowed intact followed by a tablet crushed and administered via nasogastric (NG) tube, or the reverse sequence. Because enrollment will be staggered and males and females enrolled, the randomization will be blocked (groups of 4) to minimize imbalance in assignment to the two sequences during the enrollment period, and will be used in a bidirectional fashion to balance gender, with males entering with the lowest subject numbers (#1, #2, etc.), and females with the highest subject numbers (#32, #31, etc.) in the randomization schedule. The biomedical informatics core will generate the randomization schedule. During each inpatient phase, pharmacokinetic parameters will be monitored for 36 hours. Subjects will remain in the CTRC for 24 hours after each drug administration to allow for adequate pharmacokinetic sampling. Subjects will return to the clinic on study days 2 and 9 of the study schedule for 30 and 36 hour blood samples. Subjects will then undergo a one-week washout period and then will be crossed over to the alternative mode of administration. Subjects will be discharged from the study after vital signs are checked on study days 2 and 9 of the study schedule at 36 hours, assuming the subject is hemodynamically stable.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy - defined as being free from significant cardiac, pulmonary, gastrointestinal, hepatic, biliary, renal, hematological, neurological and psychiatric disease as determined by history, physical examination and clinical laboratory test results.
2. Male or female between 18 and 40 years of age inclusive, at the time of signing the informed consent.
3. A female is eligible to enter and participate in this study if she is of:

   i. Non-child bearing potential (i.e. postmenopausal, surgically sterile, bilateral tubal ligation, or oophorectomy); or

   ii. Child bearing potential, has a negative serum pregnancy test at screening, a negative urine pregnancy test on each admission day, and certifies compliance with one of the following:
   * Complete abstinence from intercourse from 2 weeks prior to administration of the study drug, throughout the study, and 3 days after completion or premature discontinuation from the study to account for elimination of the study drug; or
   * Sterilization of monogamous male partner; or
   * Oral contraceptives if the subject has been taking them continuously for at least three months prior to the study; or
   * Any FDA approved non-hormonal intrauterine device (IUD); or
4. Within 20% of ideal body weight based on the subject's height (inches) and weight (kg).
5. Willing and able to give written informed consent prior to entering the study.

Exclusion Criteria:

1. Participated in another study within 30 days of the study period.
2. A serum sodium less than 135 mEq/L at screening or on study days 1 or 8 of the study schedule.
3. A positive urine or serum pregnancy test, or are currently breast-feeding.
4. A history of intestinal surgery or gastrointestinal disorder that may affect drug absorption.
5. Any clinically significant abnormal result on the screening blood tests, ECG, or physical exam.
6. Use of CYP3A4 inhibitors or inducers as medications, juices, or herbal supplements within 96 hours prior to the study period.
7. Use of oral or intravenous antibiotics within 14 days of the study period.
8. A current history of alcohol or drug abuse.
9. Any alcohol consumption within 24 h prior to study days 1 and 8 of the study schedule.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 29 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration-time curve from time 0 to infinity (AUC) | PK samples: from pre-dose to 36 hours
Area under the plasma drug concentration-time curve from time 0 to the last quantifiable point (AUC(0-t)) | PK samples: from pre-dose to 36 hours
Maximum plasma concentration (Cmax) | PK samples: from pre-dose to 36 hours
Time to maximal concentration (Tmax) | PK samples: pre-dose to 36 hours

CONTACTS AND LOCATIONS:
Overall Officials: J. Herbert Patterson, PharmD, Principal Investigator — University of North Caronlina - Eshelman School of Pharmacy; Elizabeth B McNeely, PharmD, Study Director — University of North Caronlina - Eshelman School of Pharmacy
Locations (1):
- University of North Carolina Healthcare, Chapel Hill, North Carolina, United States